CLINICAL TRIAL: NCT00167596
Title: Phase III Study of Usefulness of Near Infrared Spectroscopy to Optimize Tissues Perfusion and Oxygenation in Severe Sepsis
Brief Title: Near Infrared Spectroscopy (NIRS) in Severe Sepsis
Acronym: OTO-STS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: recruitment was stopped as consequence of cessation of funding (economic crisis)
Sponsor: University of Versailles (Other)
Collaborators: Hutchinson Technology Inc (Industry); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Djillali Annane, Professor in medicine, University of Versailles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05008
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Critical Illness; Severe Sepsis
Keywords: near infrared spectroscopy; tissue oxygenation; organ dysfunction; mortality
MeSH Terms: conditions — Critical Illness; Sepsis | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Early goal directed therapy based on StO2 evaluation
  Interventions: Device: Near Infrared Spectroscopy
- 2 (Active Comparator): Early goal directed therapy
  Interventions: Device: conventional

INTERVENTIONS:
Device: Near Infrared Spectroscopy — resuscitation will be based on Surviving Sepsis Campaign guidelines AND on increasing StO2 to 80% or more in at least 2 out of the 3 following sites: thenar, masseter and deltoid
  Arms: 1
Device: conventional — resuscitation will be based according to Surviving Sepsis Campaign
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the usefulness of an optimization of muscle perfusion and oxygenation, as assessed by the NIRS technique, in critically ill patients with sepsis.

DETAILED DESCRIPTION:
The systemic inflammatory response to sepsis may cause impaired tissue oxygenation that can persist despite the restoration of a normal hemodynamic profile and systemic oxygen transport.

Therefore, the assessment of tissue oxygenation and perfusion is recommended in patients with severe sepsis.

The InSpectra tissue spectrometer relies on continuous wave near infrared (NIR) technology to estimate non invasively local tissue hemoglobin oxygen saturation in tissue (% StO2). This technology had been tested in a variety of systems: standard theoretical models of light transport, isolated blood, isolated blood-perfused animal organs and healthy human volunteers with induced limb ischemia. In critical-care medicine, NIRS has also been used to evaluate muscle oxygenation in trauma resuscitation and in lower extremity and abdominal compartment syndrome. However, NIRS has been rarely utilised to measure tissue blood flow and oxygen uptake in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Two of four criteria for the systemic inflammatory response syndrome; and one of the following:

  * systolic blood pressure =< 90 mm Hg; or
  * a blood lactate concentration => 4 mmol/l; or
  * skin marbling; or
  * impaired consciousness; or
  * urine output < 30 ml/h.

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Do-not-resuscitate status
* Advanced directives restricting implementation of the protocol
* Obesity (body mass index [BMI] > 30)
* Anasarca

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2005-07; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
A combined endpoint of mortality and sequential organ failure assessment (SOFA) score increase at day 7 is the primary efficacy endpoint | Day 7

SECONDARY OUTCOMES:
duration of mechanical ventilation | from randomization to Day 28
length of the hospital stay | from randomization to Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Djillali Annane, MD, PhD, Study Chair — Raymond Poincaré Hospital, AP-HP; Olivier Nardi, MD, Study Director — Raymond Poincaré Hospital, AP-HP; Gwenhael Colin, MD, Principal Investigator — Raymond Poincaré Hospital, AP-HP
Locations (7):
- France (3):
  - Raymond Poincaré Hospital, Garches
  - Hôpital Nord AP HM, Marseille
  - CHU Tours, Tours
- Germany (2):
  - GERLACH Herwig, Berlin
  - University Hospital Rostock, Rostock
- NANAS Serafeim, Athens, Greece
- EZAVALA Elizabeth, Barcelona, Spain

REFERENCES:
- [Derived] Nardi O, Zavala E, Martin C, Nanas S, Scheeren T, Polito A, Borrat X, Annane D. Targeting skeletal muscle tissue oxygenation (StO2) in adults with severe sepsis and septic shock: a randomised controlled trial (OTO-StS Study). BMJ Open. 2018 Mar 19;8(3):e017581. doi: 10.1136/bmjopen-2017-017581. PMID 29555789